CLINICAL TRIAL: NCT07117474
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Subcutaneous Injection of HRS-9563 in Subjects With Mild Hypertension: a Randomized, Double-blind, Placebo-controlled Phase I Study.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9563-101
Record Dates: First submitted 2025-07-09; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Subjects With Mild Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group 1: Injection of HRS-9563 or placebo (Experimental)
  Interventions: Drug: HRS-9563, placebo
- Treatment group 2: Injection of HRS-9563 or placebo (Experimental)
  Interventions: Drug: HRS-9563, placebo
- Treatment group 3: Injection of HRS-9563 or placebo (Experimental)
  Interventions: Drug: HRS-9563, placebo
- Treatment group 4: Injection of HRS-9563 or placebo (Experimental)
  Interventions: Drug: HRS-9563, placebo
- Treatment group 5: Injection of HRS-9563 or placebo (Experimental)
  Interventions: Drug: HRS-9563, placebo

INTERVENTIONS:
Drug: HRS-9563, placebo — A single subcutaneous injection of HRS-9563 injection or placebo was administered

SUMMARY:
To evaluate the safety and tolerability of a single subcutaneous injection of HRS-9563 in hypertensive subjects

ELIGIBILITY:
Inclusion Criteria:

1. Males or infertile women aged 18-65 years (inclusive);
2. Body mass index in the range of 19-28 kg/m2 (inclusive);
3. Mild primary hypertension, without antihypertensive treatment, with a mean sitting systolic blood pressure ≥ 130 mmHg and ≤ 159 mmHg during screening and baseline, and a mean 24-hour ambulatory systolic blood pressure ≥ 130 mmHg during screening.

Exclusion Criteria:

1. Abnormal daily life rhythm;
2. Any blood biochemical indicator during screening or baseline did not meet the standards in the exclusion criteria;
3. Secondary hypertension;
4. Mean sitting diastolic blood pressure ≥ 100 mmHg;
5. Orthostatic hypotension;
6. History of type 2 diabetes mellitus or poorly controlled blood glucose;
7. Recently received any antihypertensive medications or medications that affect blood pressure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of any adverse events | Evaluation was performed up to Day169

SECONDARY OUTCOMES:
Maximum observed plasma concentration of HRS-9563 (Cmax) | Evaluation was performed up to Day3
Time to Cmax (Tmax) | Evaluation was performed up to Day3
Area under the concentration-time curve from 0 to the last measurable time point after HRS-9563 administration (AUC0-t) | Evaluation was performed up to Day3
Area under the concentration-time curve from time 0 to infinity after HRS-9563 administration (AUC0-inf) | Evaluation was performed up to Day3
Terminal elimination half-life of HRS-9563 (t1/2 | Evaluation was performed up to Day3
Apparent clearance of HRS-9563 (CL/F) | Evaluation was performed up to Day3
Apparent volume of distribution during terminal elimination phase of HRS-9563 (Vz/F) | Evaluation was performed up to Day3
Cumulative amount of drug excreted in urine (Ae,urine) | Evaluation was performed up to Day3
Cumulative percentage of dose recovered in urine (Fe,urine) | Evaluation was performed up to Day3

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided